CLINICAL TRIAL: NCT01011387
Title: A Prospective, Open, Non-controlled Clinical Investigation to Evaluate a NPWT (Negative Pressure Wound Therapy) System to be Used in the Treatment of Diabetic Foot Ulcers (DFUs) Including Post Amputation Wounds Associated With Diabetes.
Brief Title: Evaluation of Negative Pressure Wound Therapy in the Treatment of DFUs Incl. Post Amputation Wounds.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPWT 01
Record Dates: First submitted 2009-11-04; First posted 2009-11-11 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes; Foot Ulcers
Keywords: Diabetic foot ulcers
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPWT system (Other): Negative pressure wound therapy
  Interventions: Procedure: NPWT System; Device: NPWT system

INTERVENTIONS:
Procedure: NPWT System — Dressing change 3 times per week
Device: NPWT system — 3 dressing changes/week for maximum 4 weeks.

SUMMARY:
Primary objective

* To assess wound healing and granulation tissue formation when using the NPWT system

Secondary objectives

* To investigate the pain level at dressing removal
* To visually check exudate removal
* To investigate the ease of use for the subject and care giver when using the NPWT system

DETAILED DESCRIPTION:
The investigation is designed as a prospective, open, non-controlled clinical investigation.

Wounds to be treated under this protocol should be Diabetic foot ulcers (DFUs) or post amputation wounds associated with diabetes in hospitalized subjects or subjects treated at home. One ulcer or post amputation wound per subject will be treated for a maximum duration of 4 weeks. All subjects will receive negative pressure treatment with the NPWT system, -120 mm Hg.

In total, 10-15 subjects at two sites will be enrolled provided that they fulfill all the inclusion criteria and none of the exclusion criteria and have signed and dated a written informed consent.

The subjects will be consecutively allocated to a specific subject identification code and the recruitment will be competitive.

The primary variable wound healing and granulation tissue formation will be assessed by digital planimeter, digital photography and visual estimation.

Pain level and subject/investigator convenience will be assessed by convenience surveys.

An evaluable subject is defined as a subject completing the investigation with 4 weeks of treatment, a subject healed before 4 weeks of treatment or if the investigator judge that the wound has adequately responded on NPWT before 4 weeks and that continued treatment can be made with alternative treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic foot ulcers (DFUs) including post amputation wounds associated with diabetes suitable for Negative Pressure Wound Therapy according to the investigator's judgment
2. 1 cm2 ≤ Wound size ≤ 200 cm2
3. Male or female, 18 years and above
4. Signed Informed Consent Form
5. Subject understands the written subject Information

Exclusion Criteria:

1. Need for frequent dressing changes, i.e.<72 hours between the changes
2. Dry wounds
3. Critical ischemia (for wound healing) according to investigator's judgement
4. Malignancy in the wound and/or wound margin
5. Target ulcer previous not successfully treated with NPWT within 48 hours
6. Poorly controlled diabetes according to investigators judgement.
7. Osteomyelitis which has been left untreated
8. Infection which has been left untreated
9. Unexplored fistula
10. > 10% surface area necrotic tissue with eschar present after debridement
11. High risk for bleeding complications
12. Exposed major blood vessels, organs or nerves
13. Current or within 3 months treatment with chemotherapy or irradiation
14. Known hypersensitivity to the dressing material
15. Expected technically impossible to seal the film to maintain a vacuum for treatment
16. Expected non compliance with the Clinical Investigation Plan
17. Pregnancy
18. Subjects not suitable for the investigation according to the investigator's judgement
19. Subjects previously included in this investigation
20. Subjects included in other ongoing clinical investigation at present or during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Stansby, MD, Prof., Principal Investigator — Freeman Hospital, Newcastle upon tyne
Locations (2):
- United Kingdom (2):
  - Freeman Hospital, Newcastle upon Tyne
  - Norfolk & Norwich University Hospital, Norfolk,

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigation period: Feb 2010 - July 2010. In- and/or out-patients at two centers in UK were included in this investigation. Subjects included were 18 years and above with DFU including post amputation wounds associated with diabetes.Dressing changes were made 3 times/week for maximum 4 weeks.
Groups:
- Negative Pressure Wound Therapy System: The Avance NPWT system is intended to help promote wound healing, including drainage and removal of infectious material or other fluids, under the influence of continuous and/or intermittent negative pressure. Avance NPWT system is designed to be used for a wide range of wounds which are suitable for NPWT.
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy System
Started | 16
Completed | 10
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | NPWT System
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Wound Area.
Description: Measured by tracing of wound and measured by planimeter.
Time Frame: From baseline to maximum 4 weeks
Measure: Mean (Full Range); unit: cm2
Arm/Group | NPWT System
Number analyzed (Participants) | 16
cm2 | -33.7 [-82 to 15]

ADVERSE EVENTS:
Arm/Group | NPWT System
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NPWT System (N=16)
Further revision required fourth toe Ulceration plantar aspect (Surgical and medical procedures) | 1
Ulceration plantar aspect (Skin and subcutaneous tissue disorders) | 1
Further deterioration of wound (Skin and subcutaneous tissue disorders) | 1
VAC could not maintain suction as surrounding skin deteriorated and seal could not be maintained (Skin and subcutaneous tissue disorders) | 1
Diarrhoea+nausea (General disorders) | 1
Wound deteriorated (Skin and subcutaneous tissue disorders) | 1
Developed MRSA (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Coordinating Investigator will be the lead author for the mail (primary) publication from this Investigation. For any abstract and/or manuscript the Investigators will be given at least 14 days review time before the intended submission of the document.